CLINICAL TRIAL: NCT03054766
Title: The Randomized Double-blind Controlled Clinical Trial of Combination of Intravitreal Ranibizumab With or Without Macular Laser Photocoagulation for Macular Edema Secondary to Branch Retinal Vein Occlusion
Brief Title: Combination of Intravitreal Ranibizumab With or Without Macular Laser Photocoagulation for ME Secondary to BRVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Yu Xiaobing, M.D, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 121-2016001
Record Dates: First submitted 2017-02-05; First posted 2017-02-16 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Branch Retinal Vein Occlusion; Ranibizumab; Laser Photocoagulation
Keywords: Laser Photocoagulation; Ranibizumab; Branch Retinal Vein Occlusion; Vascular Endothecial Growth Factor
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ranibizumab only (Experimental): Sham macular laser photocoagulation treatment after third ranibizumab injection with PRN intravitreal injections of ranibizumab 0.5 mg guided by BCVA stabilization
  Interventions :Ranibizumab injection Interventions :Sham macular laser
  Interventions: Drug: Ranibizumab
- Ranibizumab combined macular laser (Experimental): Macular laser photocoagulation treatment after third ranibizumab injection with PRN intravitreal injections of ranibizumab 0.5 mg guided by BCVA stabilization
  Interventions :Ranibizumab injection Interventions :Macular laser photocoagulation
  Interventions: Procedure: Ranibizumab combined macular laser; Drug: Ranibizumab

INTERVENTIONS:
Procedure: Ranibizumab combined macular laser — subjects in one group receive both macular laser photocoagulation and ranibizumab injections but ones in the other group just received ranibizumab injection.
  Arms: Ranibizumab combined macular laser
Drug: Ranibizumab — all subjections received 3+PRN ranibizumab injections by BCVA stabilization
  Other Names: Lucentis

SUMMARY:
To investigate the efficacy of laser photocoagulation combined with ranibizumab intravitreal injection in macular edema (ME) secondary to branch retinal vein occlusion (BRVO) in long term.

DETAILED DESCRIPTION:
To investigate the efficacy of ranibizumab intravitreal injections-driven by achieving vision acuity stabilization compared to combination with laser photocoagulation in Chinese patients with visual impairment in ME due to BRVO.

The result of the trial will be used to support new therapy in the BRVO in China.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or female Chinese patients ≥ 18 years of age with BRVO
3. Visual impairment due to ME secondary to BRVO in at least one eye with BCVA score between 73 and 24 and at least 24 letters in the other eye

Exclusion Criteria:

1. Pregnant or nursing (lactating) women or women of child-bearing potential without using effective contraception
2. Stroke or myocardial infarction less than 3 months prior to screening visit
3. Renal failure or creatinine levels > 2.0 mg/dl
4. Uncontrolled hypertension
5. Active ocular infection or intraocular inflammation in any eye
6. Neovascularization of the iris or neovascular glaucoma in any eye
7. History of uveitis or vitreomacular traction in any eye
8. Treatment with any anti-angiogenic drugs within 3 months prior to baseline visit in any eye
9. Glaucoma or intraocular pressure (IOP) ≥ 24 mmHg in study eye
10. Active proliferative diabetic retinopathy in study eye
11. Use of other investigational drugs within 30 days and systemic vascular endothecial growth factor (VEGF) antagonism drugs within 6 months prior to baseline visit
12. Prior laser photocoagulation or intraocular procedure within 3 months prior to baseline in study eye
13. History of intravitreal corticosteroid treatment in phakic study eye, and in aphakic or pseudophakic within 3 months prior to screening
14. History of vitrectomy in study eye
15. Other protocol defined inclusion /exclusion criteria may apply

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
visual acuity changes | one year
  comparing the changes of visual acuity between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-bing Yu, M.D, Study Chair — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
share the results of the study,and one can send message to yuxiaobing@sina.come for information

REFERENCES:
- [Background] Pece A, Isola V, Piermarocchi S, Calori G. Efficacy and safety of anti-vascular endothelial growth factor (VEGF) therapy with intravitreal ranibizumab (Lucentis) for naive retinal vein occlusion: 1-year follow-up. Br J Ophthalmol. 2011 Jan;95(1):56-68. doi: 10.1136/bjo.2009.174060. Epub 2010 Jul 3. PMID 20601660
- [Derived] Song S, Yu X, Zhang P, Gu X, Dai H. Combination of Ranibizumab with macular laser for macular edema secondary to branch retinal vein occlusion: one-year results from a randomized controlled double-blind trial. BMC Ophthalmol. 2020 Jun 19;20(1):241. doi: 10.1186/s12886-020-01498-7. PMID 32560639